CLINICAL TRIAL: NCT05487703
Title: Tofacitinib Use in Rituximab-Experienced RA Patients
Brief Title: A Study To Describe The Use Of Tofacitinib After Use Of Rituximab In Patients With Rheumatoid Arthritis In A Real-World Setting
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921420
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Clinical characteristics: clinical characteristics of adult patients with Rheumatoid Arthritis (RA) initiating tofacitinib

SUMMARY:
This study is to characterize the use of tofacitinib after use of rituximab in patients with Rheumatoid Arthritis in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the CorEvitas RA Registry and initiated tofacitinib on or after November 2012.
* Initiate tofacitinib (defined as first ever use of tofacitinib) at Registry enrollment visit or at a Registry follow-up visit after November 2012
* Have prior use of rituximab
* Have CDAI measured at baseline and appropriate follow-up visit.

Exclusion Criteria:

* There are no exclusion criteria for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a retrospective analysis of participants data using the CorEvitas RA Registry
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Casablanca, Morocco

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921420

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with rheumatoid arthritis (RA), enrolled in CorEvitas RA Registry, initiated tofacitinib with a history of rituximab use on or after 06-Nov-2012, were included in this study.
Pre-assignment Details: Total 3190 participants were screened, out of which 2872 participants did not met the inclusion criteria and only 318 participants were included in the study.
Groups:
- Tofacitinib: Participants diagnosed with RA, enrolled in CorEvitas RA registry who initiated tofacitinib with a history of rituximab use on or after 06-Nov-2012 were included in this reporting group. Duration of data collection for this study was from 06-Nov-2012 to 31-Oct-2022 (approximately 9 years).
Period: Overall Study
Arm/Group | Tofacitinib
Started | 318
Subset With 6 Month Visit | 232
Completed | 209
Not Completed | 109
Not completed — Other | 19
Not completed — Participant not well | 5
Not completed — Insurance Reasons | 6
Not completed — Physician Decision | 19
Not completed — Lack of Efficacy | 60

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were observed in this study.
Arm/Group | Tofacitinib
Number analyzed (Participants) | 318
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 262
  Male | 56
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: "Number Analyzed" refers to number of participants, with available data for this measure.
  Participants
    number analyzed (Participants) | 314
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 277
    More than one race | 0
    Unknown or Not Reported | 37
Body Weight [Mean (Standard Deviation); unit: Kilograms] | 86.0 (22.3)
Body Mass Index (BMI) Categorical [Count of Participants; unit: Participants] — Body Mass Index (BMI) was classified as Normal or underweight which indicated participants with BMI (kg/m^2) less than 25 (<25), Overweight which indicated participants with BMI (kg/m^2) from 25 to less than 30 (25-<30) and obese which indicated participants with BMI (kg/m^2) greater than or equal to 30 (>=30). Population: "Number Analyzed" refers to number of participants, with available data for this measure.
  Participants
    number analyzed (Participants) | 314
    BMI (kg/m^2) <25 | 71
    BMI (kg/m^2) 25.0 to <30 | 74
    BMI (kg/m^2) >=30 | 169

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants According to Type of Health Insurance Plan
Description: Number of participants according to type of health insurance plan was reported in this outcome measure. The health insurance plan included private, Medicare, Medicaid and no insurance. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib. One participant might have more than one type of insurance.
Time Frame: At index date, index date could be anytime during observation period from 06-Nov-2012 to 31-Oct-2022, approximately 9 years (data was observed retrospectively in this study from 14-Nov-2022 to 23-Dec-2022, for approximately 1 month)
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Groups:
- Tofacitinib: Subset With 6-month Visit: Participants diagnosed with RA, enrolled in CorEvitas RA registry who initiated tofacitinib with a history of rituximab use on or after 06-Nov-2012 and with 6-month visit were included in this reporting group.
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Participants
  Private | 210 | 153
  Medicare | 147 | 112
  Medicaid | 20 | 15
  No Insurance | 4 | 2

2. Primary Outcome: Number of Participants With College Graduation or Higher Education
Description: Number of participants who were college graduate or had higher education were reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here ''Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 311 | 226
Participants | 206 | 152

3. Primary Outcome: Number of Participants According to Smoking Status
Description: Number of participants according to smoking status was reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 314 | 228
Participants
  Never smoker | 149 | 107
  Former smoker | 110 | 79
  Current smoker | 55 | 42

4. Primary Outcome: Number of Participants According to Work Status
Description: Number of participants according to work status was reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 310 | 226
Participants
  Full time | 84 | 65
  Part time | 19 | 14
  Work at home | 24 | 17
  Student | 1 | 1
  Disabled | 83 | 60
  Retired | 99 | 69

5. Primary Outcome: Number of Participants According to Alcohol Use
Description: Number of participants according to alcohol use were reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 301 | 222
Participants
  None/ less than (<)1 drink per week | 224 | 171
  1-3 drinks per week | 52 | 35
  1-2 drinks per day | 24 | 15
  Greater than (>) 3 drinks per day | 1 | 1

6. Primary Outcome: Number of Participants According to History of Comorbidities
Description: Number of participants according to history of comorbidities were reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib. One participant might have more than one history of comorbidities.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Participants
  Malignancy | 51 | 36
  Serious Infection | 58 | 40
  Tuberculosis (active or latent) | 2 | 1
  Cardiovascular Disease | 136 | 106
  Hypertension | 110 | 83
  Diabetes mellitus | 43 | 30
  Interstitial Lung Disease (ILD/Pulmonary Fibrosis) | 8 | 7

7. Primary Outcome: Duration of Rheumatoid Arthritis at Index Date
Description: Duration of rheumatoid arthritis in participants at the time of index date was reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Years | 17.5 (11.0) | 18.2 (11.8)

8. Primary Outcome: Age at Onset of Rheumatoid Arthritis at Index Date
Description: Participants age at onset of rheumatoid arthritis at the time of index date was reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Years | 42.3 (13.9) | 42.2 (14.4)

9. Primary Outcome: Clinical Disease Activity Index (CDAI)
Description: CDAI was a simplified index for assessing the disease activity comprising of the swollen joint counts (SJC), tender/painful joint counts (TJC), participant's global assessment of disease activity (PtGA) and physician's global assessment of disease activity (PGA). CDAI is the numerical sum of 4 outcome parameters: SJC and TJC (based on 28-joint assessment range from 0 to 28, higher scores indicated worse condition), PtGA and PGA (score range from 0 to 10, assessed on 0-10 centimeter (cm) visual analog scale (VAS); higher scores indicated greater affection due to disease activity). CDAI total score = 0 (no disease) to 76 (severe disease), higher scores indicated worse condition. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Units on a scale | 23.1 (14.7) | 22.3 (14.0)

10. Primary Outcome: Number of Participants According to CDAI Categories
Description: Number of participants according to CDAI category were reported in this outcome measures. CDAI was simplified index for assessing disease activity comprising of SJC, TJC, PtGA and PGA. CDAI is numerical sum of 4 outcome parameters: SJC and TJC (based on 28-joint assessment range from 0 to 28, higher score indicated worse condition), PtGA and PGA (score range from 0 to 10, assessed on 0-10 cm VAS; higher score indicated greater affection due to disease activity). CDAI total score = 0 (no disease) to 76 (severe disease), higher score indicated worse condition. Score range-Remission: CDAI less than or equal to (<=) 2.8. Low Disease Activity: CDAI greater than (>) 2.8 and <= 10. Moderate Disease Activity: CDAI > 10 and <= 22. High Disease Activity: CDAI > 22. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 310 | 226
Participants
  Remission (<= 2.8) | 17 | 13
  Low (> 2.8 to <=10) | 53 | 38
  Moderate (>10 to <= 22) | 84 | 64
  High (>22) | 156 | 111

11. Primary Outcome: Tender Joint Count
Description: Tender joint count was used to measure the pain and inflammation in the joints, based on 28-joint assessment range from 0 to 28, where higher scores indicated worse condition. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: Joint count
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Joint count | 8.6 (8.1) | 8.3 (7.8)

12. Primary Outcome: Swollen Joint Count
Description: Swollen joint count was used to measure the pain and inflammation in the joints. Based on 28-joint assessment range from 0 to 28, where higher scores indicated worse condition. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: Joint count
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Joint count | 5.5 (5.2) | 5.2 (5.0)

13. Primary Outcome: Patient Global Assessment (PGA) VAS
Description: PGA-VAS was used to assess disease activity; assessed on 0-100 millimeter (mm) VAS; higher scores indicated greater affection due to disease activity. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Millimeter | 52.8 (25.8) | 51.4 (25.6)

14. Primary Outcome: Modified Health Assessment Questionnaire (mHAQ)
Description: mHAQ is the modified version of HAQ which simplifies it from 20 questions to 8 questions, which assessed the ability to perform tasks due to rheumatoid arthritis. It comprised of 8 questions on 8 categories of daily living activities: dress/groom; arise; eat; grip; walk; hygiene; reach; and common activities over past week before specified time point. Eight items were rated on a 4-point Likert scale from 0 to 3, where 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total score ranged from 0 to 3, where 0 = least difficulty and 3 = extreme difficulty, higher scores indicated worse functioning. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Units on a scale | 1.3 (0.7) | 1.3 (0.7)

15. Primary Outcome: Pain VAS
Description: Pain VAS was assessed using 100 millimeter (mm) horizontal line to rate pain. Score ranged from 0 mm to 100 mm; where, 0 = no pain and 100 = worst possible pain. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Millimeter | 58.0 (27.0) | 57.1 (26.6)

16. Primary Outcome: Fatigue VAS
Description: Participants assessed their fatigue using a 0 to 100 mm VAS scale, where 0 mm = no fatigue and 100 mm = worst possible fatigue. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Millimeter | 58.3 (28.5) | 57.3 (29.1)

17. Primary Outcome: Number of Participants With European Quality of Life-5 Dimensions-3 Level (EQ-5D-3L) Domain Scores of 2 or Higher
Description: EQ-5D-3L is a health profile questionnaire used to assess quality of life along 5 dimensions. Participants rated 5 aspects of health (walking, self-care, usual activities, pain/discomfort, and anxiety/depression) by choosing from 3 answering options (1=no problems; 2=some problems; 3=extreme problems). The mean of the summed score ranged from 1 to 3 with "1" corresponding to no problems and "3" corresponding to severe problems in the 5 dimensions, where higher score indicated more severe problems. In this outcome measure number of participants with a domain score of 2 or higher in each individual domain are reported. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Participants
  Walking | 229 | 167
  Self-care | 161 | 123
  Usual activities | 232 | 173
  Pain and discomfort | 228 | 170
  Anxiety and depression | 145 | 99

18. Primary Outcome: Number of Participants According to Previous Drug Therapies With Conventional Disease-Modifying Antirheumatic Drug (csDMARD)
Description: Number of participants according to previous drug therapies with csDMARD were reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Participants
  0 previous csDMARD | 7 | 6
  1 previous csDMARD | 69 | 51
  >= 2 previous csDMARD | 242 | 175

19. Primary Outcome: Number of Participants According to Line of Therapy at Tofacitinib Initiation
Description: Number of participants were classified according to line of therapy in which Tofacitinib was initiated and were reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Participants
  2 prior biologics (Rituximab (RTX) + 1 other biologic) | 9 | 9
  3 prior biologics (RTX + 2 other biologics) | 18 | 15
  4 prior biologics (RTX + 3 other biologics) | 291 | 208

20. Primary Outcome: Number of Participants According to Concomitant Therapies
Description: Number of participants classified according to concomitant therapies were reported in this outcome measure. One participant might have received more than one concomitant therapy. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Participants
  Monotherapy | 147 | 103
  Combination with Methotrexate (MTX) only | 85 | 71
  Combination with nonMTX csDMARD only | 55 | 36
  Combination with MTX & nonMTX csDMARD | 31 | 22
  Prednisone | 112 | 81

21. Primary Outcome: Percentage of Participants Who Used Rituximab (RTX) Directly Before Tofacitinib
Description: Percentage of participants who used rituximab directly before tofacitinib were reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Percentage of participants | 36.9 | 36.4

22. Primary Outcome: Duration of Prior Rituximab (RTX) Use
Description: Duration of prior RTX use (in months) was reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Months | 23.6 (25.3) | 22.8 (24.6)

23. Primary Outcome: Number of Participants According to Line of Therapy at Rituximab Initiation
Description: Number of participants were classified according to line of therapy in which Rituximab was initiated were reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 195 | 141
Participants
  2 prior biologics (other biologic + Rituximab [RTX]) | 33 | 28
  3 prior biologics (2 other biologics + RTX) | 64 | 50
  4 prior biologics (3 other biologic + RTX) | 98 | 63

24. Primary Outcome: Number of Participants According to Year of Rituximab Discontinuations
Description: Number of participants were classified according to year of rituximab discontinuations and were reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 259 | 187
Participants
  2006-2007 | 7 | 6
  2008-2009 | 20 | 14
  2010-2011 | 42 | 30
  2012-2013 | 71 | 52
  2014-2015 | 56 | 41
  2016-2017 | 37 | 27
  2018-2019 | 18 | 11
  2020-2022 | 8 | 6

25. Primary Outcome: Percentage of Participants Who Discontinued Rituximab
Description: Percentage of participants who discontinued rituximab were reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Percentage of participants | 34.3 | 0

26. Primary Outcome: Number of Participants According to Reason for Discontinuation of Rituximab
Description: Number of participants were classified according to reasons for discontinuation of rituximab and were reported in this outcome measure. Reasons for discontinuation of rituximab included safety, effectiveness, insurance, participant doing well and other reasons. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here ''Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure. This outcome measure was planned to be analyzed only in tofacitinib group.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 109
Participants
  Effectiveness | 60
  Physician Decision | 19
  Insurance | 6
  Participant doing well | 5
  Other Reasons | 19

27. Primary Outcome: Number of Participants According to Tofacitinib Initiation Year
Description: Number of participants were classified according to year of tofacitinib initiation and were reported in this outcome measure. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 318 | 232
Participants
  2012-2013 | 81 | 62
  2014-2015 | 80 | 56
  2016-2017 | 83 | 63
  2018-2019 | 49 | 34
  2020-2022 | 25 | 17

28. Primary Outcome: Change From Baseline in CDAI at 6 Months Follow-up
Description: CDAI was a simplified index for assessing the disease activity comprising of the swollen joint counts (SJC), tender/painful joint counts (TJC), participant's global assessment of disease activity (PtGA) and physician's global assessment of disease activity (PGA). CDAI is the numerical sum of 4 outcome parameters: SJC and TJC (based on 28-joint assessment range from 0 to 28, higher scores indicated worse condition), PtGA and PGA (score range from 0 to 10, assessed on 0-10 centimeter (cm) visual analog scale; higher scores indicated greater affection due to disease activity). CDAI total score = 0 (no disease) to 76 (severe disease), higher scores indicated worse condition. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: Baseline, Month 6 follow up visit (anytime during observation period from 06-Nov-2012 to 31-Oct-2022, approximately 9 years [data was observed retrospectively in this study from 14-Nov-2022 to 23-Dec-2022, for approximately 1 month])
Population: Analysis population included all eligible participants whose medical records were retrieved, observed in this study and who had completed 6-month follow up visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 232
Units on a scale
  At baseline | 22.53 (14.04)
  At 6 Months | 19.08 (14.02)

29. Secondary Outcome: Percentage of Participants Who Achieved Minimum Clinically Important Difference (MCID) at 6 Month Follow Up
Description: MCID improvement was assessed based on health assessment questionnaire (HAQ). HAQ: self-reported, valid assessment of functional disability in RA. Assessed based on ability of participants to perform daily activities in 8 categories: dressing, arising, eating, walking, reaching, gripping, hygiene, and conducting daily activities. Eight items were rated on a 4-point Likert scale from 0 to 3, where 0= without any difficulty, 1= with some difficulty, 2= with much difficulty, and 3= unable to do. Overall score was computed as sum of domain scores and divided by number of domains answered. Total score ranged from 0 to 3, where 0= least difficulty and 3= extreme difficulty, higher scores indicating worse functioning. Achievement of MCID for HAQ was defined as decrease in minimum of 0.22 units from baseline. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 232
Percentage of participants | 28.6 [22.7 to 35.2]

30. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) at 6 Months Follow-up
Description: HAQ: self-reported, valid assessment of functional disability in RA. The 20-question instrument assessed ability of participants to perform daily activities in 8 functional areas: dressing, arising, eating, walking, hygiene, reaching, griping, and conducting daily activities. Eight items were rated on a 4-point Likert scale from 0 to 3, where 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total score ranged from 0 to 3, where 0 = least difficulty and 3 = extreme difficulty, higher scores indicating worse functioning. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 232
Units on a scale
  At baseline | 1.35 (0.67)
  At 6 Months | 1.28 (0.68)

31. Secondary Outcome: Change From Baseline in Pain VAS at 6 Months Follow-up
Description: Pain VAS was assessed using 100 mm horizontal line to rate pain. Score ranged from 0 mm to 100 mm; where, 0 = no pain and 100 = worst possible pain. Index date was defined as the date of tofacitinib initiation at or after enrollment in the registry; initiation was defined as first ever use of tofacitinib.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 232
Units on a scale
  At baseline | 57.16 (26.74)
  At 6 Months | 51.27 (27.80)

32. Secondary Outcome: Change From Baseline in Fatigue VAS at 6 Months Follow-up
Description: as for outcome 16
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib: Subset With 6-month Visit
Number analyzed (Participants) | 232
Units on a scale
  At baseline | 57.39 (29.19)
  At 6 Months | 54.75 (29.30)

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not planned to be collected during the study.
Description: Minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not be met. Hence, adverse events were not collected and reported.
Arm/Group | Tofacitinib | Tofacitinib: Subset With 6-month Visit
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT05487703/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT05487703/SAP_001.pdf